CLINICAL TRIAL: NCT06987227
Title: Effects of a Smart Parent-child Bonding Intervention on the Physical, Psychological, and Social Health of Parents of Preterm Infants During Hospitalization and Home Return: a Randomized Controlled Trial
Brief Title: Effects of Intelligent Parent-child Bonding Intervention on the Physical, Psychological and Social Health of Parents of Premature Infants During Hospitalization and Return Home
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Defense Medical Center, Taiwan (Other)
Responsible Party: Principal Investigator, Hsiang-Yun Lan, Associate Professor, National Defense Medical Center, Taiwan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: B2025050055
Record Dates: First submitted 2025-04-18; First posted 2025-05-23 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-04

CONDITIONS: Parents of Premature Infants; Intelligent Intervention; Parent-child Connection
Keywords: physical health; psychological health; parents of premature infants; social health; Intelligent intervention; parent-child connection
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intelligent intervention to enhance parent-child connection (Experimental): In addition to routine care, premature infants will receive "intelligent parent-child connection intervention" during hospitalization and continue to use it until one month after the premature infant returns home.
  Interventions: Behavioral: Intelligent intervention to enhance parent-child connection; Other: Routine care
- Routine care group (Active Comparator): Routine care is provided to premature infants during hospitalization, and general nursing guidance for premature infant discharge care is provided before discharge.
  Interventions: Other: Routine care

INTERVENTIONS:
Behavioral: Intelligent intervention to enhance parent-child connection — The "Intelligent Intervention to Enhance Parent-Child Connection" support program is mainly carried out through web pages, Figma software, cloud files and official Line accounts. It can be divided into: the first stage is to provide parents with care knowledge and skills during the hospitalization of premature infants, provide parents with physical and mental support, and encourage parents to establish parent-child connections and prepare for discharge. The second stage is after discharge, continuing to provide premature infants' families with the care guidance needed to respond to the different stages of development of premature infants, including interpersonal support, sleep schedule establishment, crying comfort, premature infant nutrition and couple relationship management, etc., and continue to provide family support, answer questions and track its implementation status.
  Arms: Intelligent intervention to enhance parent-child connection
Other: Routine care — Premature infants receive routine care during their hospitalization, and general nursing guidance for premature infant discharge care is provided before discharge.

SUMMARY:
The study purpose is to construct and validate the effects of "intelligent parent-child bonding intervention" on the physical, psychological and social health of parents of premature infants.

DETAILED DESCRIPTION:
Background:

Premature babies are born at 20 weeks but less than 37 weeks of gestation. In 2020, there were approximately 13.4 million premature babies worldwide, accounting for 10% of the total number of newborns. Although Taiwan's birth rate has declined, the premature birth rate has increased year by year due to factors such as late marriage and childbirth at an advanced age, reaching 10.88% in 2023. Premature birth survivors face long-term physical and psychological challenges that affect their quality of life and cause significant stress for their families, including anxiety and depression. Mother-child separation is considered "toxic stress" that affects parent-child relationships and family function. Therefore, establishing a bond with your newborn is critical to the health of both the parents and the premature infant.

Methods:

This study was a three-year randomized controlled trial using a longitudinal repeated measures design. Convenience sampling will be used to recruit 360 parents of premature infants in the pediatric and neonatal intensive care unit of a northern medical center. Participants will be randomly assigned to two conditions (usual care and smart parent-child bonding intervention). The intervention will begin during the premature infant's hospital stay until the first month after discharge. Data will be collected using questionnaires and biometrics. Outcome variables included sleep status, fatigue, stress, anxiety, depression, self-efficacy, parent-child connection, partner relationship, family resilience, and quality of life of parents of preterm infants. In addition, these data will be collected before the intervention, 2 weeks after the intervention, before premature infants are discharged from the hospital, and in the first month after premature infants return home. It is expected that the generalized estimating equation method will be used to analyze the research results.

ELIGIBILITY:
Inclusion Criteria: 1. Parents of premature infants born less than 37 weeks of age; 2. Parents of premature infants aged 20 or above and able to communicate in Mandarin and Taiwanese; 3. Parents of premature infants agree to participate in this study and sign the research consent form; 4. The child is currently in the Pediatric and Neonatal Intensive Care Center

Exclusion Criteria: 1. The premature baby has congenital abnormalities or is in critical condition and cannot survive; 2. The parents cannot use mobile phones or other Internet devices; 3. The parents have a history of mental illness, intellectual disability or substance abuse.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2025-06-15 (Estimated); Primary Completion 2028-03-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
The Pittsburgh Sleep Quality Index, PSQI | Changes in parents' sleep patterns before premature infants are discharged from hospital and in the first month after premature infants return home
  The sleep quality in the past month was measured, including seven indicators: subjective statement of sleep quality, sleep latency, sleep duration, sleep efficiency, sleep disturbance, use of sleep aids and daytime dysfunction. Each indicator was scored between 0-3 points, and the total score ranged from 0-21 points. The higher the score, the worse the sleep quality. When the total score of sleep quality is >5 points, it means poor sleep quality, and the total score of sleep quality is ≤5 points, it means good sleep quality.
Actigraphy and Sleep Diary measures sleep details | Changes in parents' sleep details before premature infants are discharged from hospital and in the first month after premature infants return home
  The Cole-Kripke algorithm was used to calculate the following data: (1) total sleep time: the actual time of falling asleep; (2) sleep efficiency: the percentage of time in bed compared to the actual sleep time; (3) sleep latency: the time from the time in bed to the time of falling asleep recorded by the actigraph; and (4) number of awakenings: the number of awakenings during a sleep cycle. The sleep log is recalled by the primary caregiver immediately after waking up every day, recording the sleep time and sleep status of the previous day, in order to understand the total sleep hours, the number of awakening hours/times at night, sleep efficiency, and whether there are any events that affect the mood for falling asleep, medication or physical discomfort, whether stimulants and alcohol are consumed, etc., and the sleep quality of the previous night and the degree of wakefulness when waking up are evaluated on a scale of 1 to 5 points.
Brief Fatigue Inventory, BFI | Changes in parental fatigue before premature infants were discharged from hospital and in the first month after they returned home
  The scale is divided into two parts: the severity of fatigue and the degree of interference of fatigue on life. There are 9 questions in total, each with a score of 0 to 10 points. The total score is calculated as the average score of the first part plus the average score of the second part. The higher the score, the higher the degree of fatigue.
Perceived Stress Scale, PSS | Changes in parental perceived stress before premature infants were discharged from hospital and in the first month after they returned home
  This scale is used to measure the stress level in an individual's life. The original scale has 14 questions, using the Likert scoring method, with a scoring method ranging from 0 (never), 1 (occasionally), 2 (sometimes), 3 (often) to 4 (always). Questions 4, 5, 6, 7, 9, 10, and 13 are reverse scored. The total score ranges from 0 to 56. The higher the score, the higher the stress level of the subject.
Postpartum Specific Anxiety Scale | Changes in parental anxiety before premature infants were discharged from hospital and in the first month after they returned home
  The frequency scale used to assess the anxiety focused on mothers and infants experienced by women in the past week has a total of 12 questions, which are classified into four sub-items according to the content: maternal ability and attachment anxiety, infant safety and health anxiety, infant care anxiety, and maternal psychosocial adaptation. The Likert four-point scoring method is used, with each question ranging from 1 to 4 points, from low to high representing "never", "rarely", "often", and "always". The total score ranges from 12 to 48 points, and the higher the score, the higher the level of anxiety.
Edinburgh Postpartum Depression Scale | Changes in parental depression before premature infants were discharged from hospital and in the first month after they returned home
  There are 10 questions in total. Each item is scored from 0 to 3 points, and the total score range is 0 to 30 points. The higher the score, the more severe the depression symptoms. It is recommended that scores of ≧10 and ≧9 be used as the criteria for screening postpartum depression symptoms for fathers and mothers respectively.
Parental Self-efficacy scale, PSE Scale | Changes in parental self-efficacy before premature infants were discharged from hospital and in the first month after they returned home
  It is divided into three aspects: (1) Parenting role evaluation: refers to the overall feeling of one's own parenting effectiveness; (2) Parenting confidence: refers to the feeling of whether one has the confidence and competence to do the work of raising children; (3) Parenting ability: refers to the recognition and understanding of one's own ability to actually carry out the work of raising children. The scale has 20 questions, which are scored on a Likert scale, with a total score of 20-100 points. The higher the score, the higher the evaluation of one's own parenting ability. There are seven questions about parenting confidence, all of which are reverse questions.
Parent-infant bonding | Changes in parent-infant bonding before premature infants were discharged from hospital and in the first month after they returned home
  The scale questions adopt the Likert six-point scoring method, with each question scoring from 1 to 6 points, and the options range from "strongly disagree" to "strongly agree". Among them, only the "parenting adaptation" item adopts the reverse scoring method. The higher the score, the better the mother-infant connection in this dimension.
Relationship Assessment Scale, RAS | Changes in parental relationship before premature infants were discharged from hospital and in the first month after they returned home
  The scale consists of 7 questions, using the Likert five-point scoring method. Each question has a score of 1 to 5. The number 1 indicates the lowest score (such as "very poor" or "unsatisfied"), and the number 5 indicates the highest score (such as "very good" or "completely satisfied"). Please answer according to your own feelings. The total score ranges from 7 to 35 points. The higher the score, the more satisfied the individual is with the relationship between husband and wife/partner.
Family Resilience Assessment | Changes in family resilience before premature infants were discharged from hospital and in the first month after they returned home
  This scale has a total of 31 questions, covering three categories, namely belief system (a total of 13 questions), organizational model (a total of 9 questions) and family communication process (a total of 9 questions). It adopts Likert's five-point scoring method, "strongly agree" (5 points) and "strongly disagree" (1 point). The higher the score, the better the family resilience.
World Health Organization Quality of Life-BREF, WHOQOL-BREF | Changes in quality of life before premature infants were discharged from hospital and in the first month after they returned home
  There are 28 questions in total, with the past two weeks as the reference point, to assess the quality of life. The content includes four aspects: physical health, psychology, social relations and environment. The Likert five-point scoring method is adopted. The higher the score, the better the quality of life.

IPD SHARING:
Plan to Share IPD: No